CLINICAL TRIAL: NCT03712917
Title: Comparison of Therapeutic Effects of Greater Occipital Nerve Block, Topiramate, and Flunarizine on Episodic Migraine: A Randomised Parallel Group Study
Brief Title: Comparison of Therapeutic Effects of Greater Occipital Nerve Block, Topiramate, and Flunarizine on Episodic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mustafa Ceylan, Principal İnvastigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/22-3
Record Dates: First submitted 2018-10-13; First posted 2018-10-19 (Actual); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Migraine
Keywords: Migraine; Greater Occipital Nerve Block; Topiramate; Flunarizine
MeSH Terms: conditions — Migraine Disorders | interventions — Topiramate; Flunarizine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Greater Occipital Nerve Block (Active Comparator): The GONB solution is prepared with 1 ml triamcinolone (40mg), 2 ml bupivacaine (10 mg), and 1 ml 0,9% NaCl. The solution is administered using a 22G × 1¼" (0.7 × 40mm) injector with the patient lying prone on the table. Injection is applied to medial of the occipital artery localized at the medial one-third of the superior nuchal line between the occipital tubercle and mastoid process. The scalp is cleaned with iodine before the procedure, and the injections are performed bilaterally at a volume of 2 mL after negative aspiration for blood.
  Interventions: Procedure: Greater Occipital Nerve Block
- Topiramate (Active Comparator): Topiramate is administered twice a day at a dose of 25 mg/day, which is increased to 100 mg/day in the second week.
  Interventions: Drug: Topiramate
- Flunarizine (Active Comparator): Flunarizine is introduced with a single dose of 10 mg/day.
  Interventions: Drug: Flunarizine

INTERVENTIONS:
Procedure: Greater Occipital Nerve Block — An enjection to paralyze the occipital nerve.
  Arms: Greater Occipital Nerve Block
Drug: Topiramate — An antiepileptic agent used for migraine prophylaxis.
  Arms: Topiramate
Drug: Flunarizine — A calcium overload blocker agent used for migraine prophylaxis.
  Arms: Flunarizine

SUMMARY:
Background: Preventive drug therapy in migraine aims to reduce the attack frequency, severity and duration of headache. Flunarizine and topiramate are widely used in the prevention of migraine attacks. Greater occipital nerve block (GONB) is an alternative treatment option for the prophylactic treatment of migraine. In this study, investigators compared the effectiveness of GONB, topiramate, and flunarizine in terms of reduction in post-treatment VAS scores and attack frequencies in patients with episodic migraine in a four-week period.

Material and Methods: At least one hundred and twenty migraine patients are aimed to be randomly divided into three treatment groups, namely flunarizine (n=40, estimated), topiramate (n=40, estimated) and GONB (n=40, estimated). The patients will be followed up for four weeks and the attack frequencies and VAS scores will be recorded weekly. At the end of the fourth week, the response rates based on 50% and 75% or more reduction in the VAS scores and attack frequencies will be calculated. Group-wise comparisons will be assessed statistically.

ELIGIBILITY:
Inclusion Criteria:

1. Migraine diagnosis according to ICHD-2
2. Ages between 15 -45 Volunteering
3. Monthly attack number between 5-14
4. BMI between 18-30
5. w/o history of nephrolithiasis
6. w/o history of DM, peripheral vascular disease
7. w/o history of chronic systemic diseases (lung, heart,liver, kidney)
8. w/o any detected CNS disease (including MS, movement disorders, CVD, primary or secondary tumors)
9. w/o history of acute or chronic psychiatric disease
10. w/o history of antiplatelet and anticoagulant medication
11. w/o any combination of medication overuse headache or other primary headaches
12. w/o previous medication of flunarizine and topiramate
13. w/o previous application of GONB

Exclusion Criteria:

1. Pregnancy
2. Lost to follow up

   * exited with his/her own will
   * detected primary headache during follow up
   * cessation due to adverse effects of topiramate
   * cessation due to adverse effects of flunarizine

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Resarch Hospital, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diener H-C, Goadsby PJ. Migraine In: Brandt T, Caplan L, Dichgans J, Diener H-C, Kennard C (eds) Course and treatment of neurological disorders. 2nd edition. Academic Press, San Diego, (2003). pp 1-16.
- [Background] Baker C. Double-blind evaluation of flunarizine and placebo in the prophylactic treatment of migraine. Headache 1987; 27:288.
- [Background] Silberstein SD, Neto W, Schmitt J, Jacobs D; MIGR-001 Study Group. Topiramate in migraine prevention: results of a large controlled trial. Arch Neurol. 2004 Apr;61(4):490-5. doi: 10.1001/archneur.61.4.490. PMID 15096395
- [Background] Bovim G, Sand T. Cervicogenic headache, migraine without aura and tension-type headache. Diagnostic blockade of greater occipital and supra-orbital nerves. Pain. 1992 Oct;51(1):43-48. doi: 10.1016/0304-3959(92)90007-X. PMID 1454403

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Greater Occipital Nerve Block | Topiramate | Flunarizine
Started | 40 | 40 | 40
Completed | 31 | 32 | 31
Not Completed | 9 | 8 | 9
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Adverse Event | 0 | 4 | 3
Not completed — Lost to Follow-up | 9 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Greater Occipital Nerve Block | Topiramate | Flunarizine | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Row population is the defined after the exclusion of patients from overall study population
  years
    number analyzed (Participants) | 31 | 32 | 31 | 94
    (all) | 30.2 (8.9) | 31.5 (8.2) | 30.9 (9.0) | 30.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Row population is the defined after the exclusion of patients from overall study population
  Participants
    number analyzed (Participants) | 31 | 32 | 31 | 94
    Female | 22 | 26 | 24 | 72
    Male | 9 | 6 | 7 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 40 | 40 | 40 | 120
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale
Description: Range Pain 0-10, 0: No pain, 10: Worst Pain
Time Frame: Post treatment 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Greater Occipital Nerve Block | Topiramate | Flunarizine
Number analyzed (Participants) | 31 | 32 | 31
score on a scale
  Pretreatment | 8.1 (1.0) | 7.9 (0.9) | 7.9 (0.9)
  Posttreatment | 5.9 (1.6) | 5.5 (2.1) | 5.3 (1.7)

2. Primary Outcome: Attack Frequencies
Description: Number of headaches patients suffer in a month.
Time Frame: Post treatment 4 weeks
Measure: Mean (Standard Deviation); unit: headaches per month
Arm/Group | Greater Occipital Nerve Block | Topiramate | Flunarizine
Number analyzed (Participants) | 31 | 32 | 31
headaches per month
  Pretreatment | 8.6 (2.6) | 8.0 (2.7) | 8.0 (2.4)
  Posttreatment | 3.3 (1.0) | 2.7 (2.3) | 2.8 (1.4)

ADVERSE EVENTS:
Time Frame: From the start of the study till the end (one month)
Arm/Group | Greater Occipital Nerve Block | Topiramate | Flunarizine
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 4/40 | 3/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Greater Occipital Nerve Block (N=40) | Topiramate (N=40) | Flunarizine (N=40)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) — Mild daytime sedation
Fatique (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
memory difficulties (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT03712917/Prot_SAP_000.pdf